CLINICAL TRIAL: NCT05412472
Title: A Phase 1, Open-Label, Single-Dose, Parallel-Group Study to Evaluate the Effects of Renal Impairment on the Pharmacokinetics, Safety and Tolerability of GC4419
Brief Title: Study to Evaluate the Effects of Renal Impairment on the Pharmacokinetics, Safety and Tolerability of GC4419
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTI-4419-003
Record Dates: First submitted 2022-06-07; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — avasopasem manganese

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 1) Healthy subjects with normal renal function (Experimental)
  Interventions: Drug: GC4419
- 2) Mild renal impairment (Experimental)
  Interventions: Drug: GC4419
- 3) Moderate renal impairment (Experimental)
  Interventions: Drug: GC4419
- 4) Severe renal impairment (Experimental)
  Interventions: Drug: GC4419

INTERVENTIONS:
Drug: GC4419 — 45 mg IV infusion of GC4419 over 60 minutes.

SUMMARY:
The study is a two-center, Phase 1, open-label, single-dose, one-period, four groups, PK study in subjects with various severities of renal impairment and matched healthy controls.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in Arm 1:

1. Male or female, non-smoker ≥ 18 and ≤ 80 years of age, with BMI ≥ 18.0 and ≤ 40.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Healthy as defined by the absence of clinically significant illness and surgery within 4 weeks prior to dosing; the absence of clinically significant medical history
3. Females of childbearing potential partner must be willing to use an acceptable contraceptive method throughout the study and for 30 days after the study drug administration:
4. Male subjects who are sexually active must be willing to use one of an acceptable contraceptive method from the first dosing until at least 90 days after the study drug administration:
5. Male subjects with a pregnant partner must agree to use a condom from the first dosing until at least 90 days after the study drug administration.
6. Male subjects must be willing not to donate sperm until 90 days following study drug administration. Female subjects must avoid oocyte donation until 90 days following study drug administration.

Subjects must meet all of the following criteria to be included in Arms 2 to 4:

1. Male or female, non-smoker and/or light smoker, ≥18 and ≤80 years of age, with BMI ≥ 18.0 and ≤ 40.0 kg/m2 and body weight ≥ 50.0 kg for males and ≥ 45.0 kg for females.
2. Have a diagnosis of renal impairment that has been stable, without any significant change in overall disease status in the last 3 months
3. Have an eGFR (MDRD4 equation) at screening within the range of:

   1. Group 2 - Mild Group: 60 - 89 mL/min/1.73 m2;
   2. Group 3 - Moderate Group: 30 - 59 mL/min/1.73 m2;
   3. Group 4 - Severe Group: < 30 mL/min/1.73 m2 not requiring dialysis.
4. The absence of clinically unstable neurological, cardiovascular, pulmonary, hematological, psychiatric, or gastrointestinal illness
5. Subject may have stable treated medical illnesses and underlying diseases producing the renal impairment
6. Have normal or non-clinically significant findings at physical examination
7. Stable medical regimen deemed not to interact with study drug PK, with no changes for at least 14 days prior to dosing
8. Females of childbearing potential partner must be willing to use an acceptable contraceptive method throughout the study and for 30 days after the study drug administration:
9. Male subjects who are sexually active must be willing to use one of an acceptable contraceptive method from the first dosing until at least 90 days after the study drug administration:
10. Male subjects with a pregnant partner must agree to use a condom from the first dosing until at least 90 days after the study drug administration.
11. Male subjects must be willing not to donate sperm until 90 days following study drug administration. Female subjects must avoid oocyte donation until 90 days following study drug administration.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from Arm 1:

1. Any clinically significant abnormality at physical examination or clinically significant abnormal laboratory test results at screening.
2. Positive test for hepatitis B, hepatitis C, or HIV at screening;
3. History of anaphylaxis, hypersensitivity reaction, or a clinically significant reaction to any drug.
4. Clinically significant ECG abnormalities or vital sign abnormalities
5. History of significant alcohol abuse within one year prior to screening or regular use of alcohol within six months prior to the screening visit
6. History of significant drug abuse within one year prior to screening or use of soft drugs within 3 months prior to the screening visit or hard drugs within 1 year prior to screening
7. Participation in a clinical research study within 30 days prior to the first dosing, administration of a biological product in the context of a clinical research study within 90 days prior to the first dosing
8. Positive urine drug screen, alcohol breath test, or urine cotinine test at screening.
9. Female subject with positive pregnancy test at screening.
10. Breast-feeding or pregnant subject within 6 months prior to study drug administration.
11. Use of medication other than topical products without significant systemic absorption and hormonal contraceptives:

    1. Prescription medication within 14 days prior to dosing;
    2. Over-the-counter products and natural health products within 7 days prior to dosing
    3. A depot injection or an implant of any drug within 3 months prior to dosing.
12. Donation of plasma within 7 days prior to dosing.
13. Inability to be venipunctured and/or tolerate catheter venous access.
14. History of myasthenia gravis or carotid sinus sensitivity.

Subjects to whom any of the following applies will be excluded from Arms 2 to 4:

1. Any clinically significant abnormality at physical examination or clinically significant abnormal laboratory test results found during medical screening.
2. Positive HIV at screening.
3. Female subjects with positive pregnancy test at screening.
4. Clinically significant unstable medical conditions or clinically significant acute exacerbation of hepatic disease within 28 days of study drug administration
5. Clinically significant abnormalities
6. Clinically significant findings on ECG
7. Presence of hepatocellular carcinoma or acute hepatic disease from infection or drug toxicity.
8. Presence of clinically active stage 3 or stage 4 hepatic encephalopathy.
9. Presence of surgically-created or transjugular intrahepatic portal systemic shunts.
10. Subjects with a positive urine drug screen or alcohol test at screening.
11. Systolic blood pressure lower than 90 or over 160 mmHg, diastolic blood pressure lower than 40 or over 105 mmHg, or heart rate less than 45 or over 100 bpm at screening.
12. History of significant drug or alcohol abuse within 6 months prior to screening.
13. Participation in another clinical study within 30 days prior to dosing.
14. Use of contraindicated medications
15. Donation of plasma within 7 days prior to dosing.
16. Breast-feeding subject.
17. Inability to be venipunctured and/or tolerate catheter venous access.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-04-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profile for GC4419 (in plasma): AUC0-t | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): AUC0-inf | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): Cmax | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): Residual Area | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): Tmax | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): T1/2el | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): Kel | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): CL/F | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.
Pharmacokinetic (PK) profile for GC4419 (in plasma): Vd/F | Within 1 hour before the start of infusion and 0.5, 1 (immediately before the start of the IV line flushing process), 1.5, 2, 3, 4, 6, 8, 12, 16, 24, and 36 hours after start of infusion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Inventiv Health Clinical -Research Pharmacy Unit, Miami, Florida
  - University of Miami Division of Clinical Pharmacology, Miami, Florida

IPD SHARING:
Plan to Share IPD: No